CLINICAL TRIAL: NCT02980796
Title: The Influence of Acute Bouts of Aerobic Exercise on Neuroplasticity and Motor Learning After Stroke
Brief Title: The Influence of Exercise on Neuroplasticity and Motor Learning After Stroke
Acronym: EX-ML3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lara Boyd, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H16-01945
Record Dates: First submitted 2016-11-28; First posted 2016-12-02 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Stroke; Exercise; Rest
Keywords: Brain; MRI; Exercise; Rehabilitation; TMS
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise + practice (Experimental): Individuals will complete 20 minutes of exercise on a recumbent bicycle before practicing a novel motor task.
  Interventions: Behavioral: Exercise; Behavioral: Practice
- Rest + practice (Active Comparator): Individuals will rest for 20 minutes before practicing a novel motor task. Attention will be controlled during this time.
  Interventions: Behavioral: Practice

INTERVENTIONS:
Behavioral: Exercise — Each experimental day participants will complete an acute bout of exercise on a recumbent bike.
  Arms: Exercise + practice
Behavioral: Practice — Each experimental day participants will complete a session of skilled motor practice.

SUMMARY:
Participants will complete 11 sessions. These include screening, 5 sessions where exercise or rest (according to group assignment) are paired with practice of a motor task, MRI and Transcranial Magnetic Stimulation (TMS) before and after the intervention will be used to assess neuroplasticity (ability for the brain to reorganize and create new connections).

DETAILED DESCRIPTION:
All participants will complete baseline sessions: 1) sub-maximal exercise test to ensure safe participation in aerobic exercise (testing session [s] 1); and 2) magnetic resonance imaging (MRI) to assess brain structure and function, and 3) clinical assessments of motor function and activity. The MRI and clinical tests will be completed on s2. Between the exercise test and MRI sessions individuals will wear accelerometers for 3 days to index usual activity levels. A custom computer program will then assign participants quasi-randomly to either the rest or exercise groups stratified on age, sex, and baseline motor function. Cortical excitability will be assessed before and after either a single session of priming aerobic exercise, or rest, by group (s3). Next, priming exercise will be paired with skilled motor practice for 5 sessions (s4-8). Practice sessions will be separated by 48 hours. Importantly motor learning will be assessed via delayed, no-exercise retention tests 24-hours (s9) and 30-days (s11) after the last practice session. Activity levels (3 day accelerometry), TMS and MRI measures will be re-assessed after the second retention test (s10).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40 - 85
* Had a stroke at least 12 months ago
* OR are a healthy adult who does not have a history of neurodegenerative disorders
* Have the ability to understand English

Exclusion Criteria:

* Contraindication to brain stimulation (such as a history of seizure or epilepsy)
* Contraindication to MRI (such as a pacemaker, metal in the eyes / brain or fear of enclosed spaces)
* Neurodegenerative disorder ( such as Parkinson disease, Alzheimers disease or Multiple Sclerosis)
* Contraindications to exercise

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change response time during a novel motor task. | Baseline, After Intervention (2 weeks), 30-day follow-up
  Serial targeting task
Wolf Motor Function Task Rate | Baseline, After Intervention (2 weeks), 30-day follow-up
  Standardized test of arm motor function

SECONDARY OUTCOMES:
Transcallosal Inhibition | Baseline, After Intervention (2 weeks), 30-day follow-up
  Ipsilateral silent period
Arm Use Ratio | Baseline, After Intervention (2 weeks), 30-day follow-up
  Accelerometry
Functional magnetic resonance imaging (fMRI) | Baseline, After Intervention (2 weeks), 30-day follow-up
  Resting state fMRI
Structural magnetic resonance imaging - myelin | Baseline, After Intervention (2 weeks), 30-day follow-up
  Myelin water fraction
Structural magnetic resonance imaging - diffusion | Baseline, After Intervention (2 weeks), 30-day follow-up
  Diffusion weighted fractional anisotrophy

CONTACTS AND LOCATIONS:
Overall Officials: Lara Boyd, Pt, PhD, Principal Investigator — Univeristy of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300